CLINICAL TRIAL: NCT01877642
Title: ADASUVE®-Lorazepam Drug-Drug Interaction Study
Brief Title: ADASUVE-Lorazepam Drug-Drug Interaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AMDC-204-402
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2013-07

CONDITIONS: Healthy Volunteers
Keywords: ADASUVE; inhaled loxapine; drug drug interaction; lorazepam; acute treatment of agitation
MeSH Terms: interventions — Lorazepam; Loxapine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Open Label (lorazepam 1 mg + Inhaled loxapine 10 mg) (Other): Inhaled Staccato loxapine 10 mg + IM lorazepam 1 mg to confirm tolerability of combined treatment
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg
- Treatment Sequence ABC (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM
- Treatment Sequence ACB (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM
- Treatment Sequence BCA (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM
- Treatment Sequence BAC (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM
- Treatment Sequence CAB (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM
- Treatment Sequence CBA (Other): Treatment: A = Lorazepam 1 mg IM + inhaled placebo, B = Lorazepam 1 mg IM + inhaled loxapine 10 mg, C= Placebo IM + inhaled loxapine 10 mg
  Interventions: Drug: Lorazepam 1 mg IM; Drug: Inhaled loxapine 10 mg; Drug: Inhaled Placebo; Drug: Placebo IM

INTERVENTIONS:
Drug: Lorazepam 1 mg IM — Lorazepam 1 mg intramuscular
  Other Names: Ativan 1 mg IM
Drug: Inhaled loxapine 10 mg — Inhaled Staccato loxapine 10 mg
  Other Names: ADASUVE 10 mg
Drug: Inhaled Placebo — Inhaler with no drug in it to mimic the ADASUVE inhaler
  Other Names: Staccato Placebo
  Arms: Treatment Sequence ABC; Treatment Sequence ACB; Treatment Sequence BAC; Treatment Sequence BCA; Treatment Sequence CAB; Treatment Sequence CBA
Drug: Placebo IM — intramuscular placebo to mimic lorazepam 1 mg IM
  Other Names: Saline
  Arms: Treatment Sequence ABC; Treatment Sequence ACB; Treatment Sequence BAC; Treatment Sequence BCA; Treatment Sequence CAB; Treatment Sequence CBA

SUMMARY:
This study will compare the safety and effects over time for giving both ADASUVE and lorazepam (intramuscular) compared to that of each agent given alone.

DETAILED DESCRIPTION:
The objective of this study is to compare the safety and pharmacodynamic profiles of concomitant administration of a single dose of ADASUVE and lorazepam (IM) compared to that of each agent administered alone. Respiratory pharmacodynamics will be monitored through recordings of respirations/minute and pulse oximetry. Other pharmacodynamic safety measures will include effects on blood pressure, heart rate, sedation and psychomotor measures of attention, information processing speed, reaction time, and coordination.

Initially, 4 subjects will receive lorazepam 1 mg IM + ADASUVE 10 mg open label to validate the dose regimen. After the safety data are reviewed and the dose regimen confirmed, 18 non-obese, healthy male or female volunteers between the ages of 18 and 50 will be enrolled in this double-blinded, double-dummy, randomized, 3-period cross-over drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 50 years, inclusive.
* Body mass index (BMI) ≥18 and ≤32.
* Subjects who are willing and able to comply with the study schedule and requirements, and stay at the CRU for 9 days.
* Subjects who speak, read, and understand English and are willing and able to provide written informed consent on an IRB approved form prior to the initiation of any study procedures.
* Subjects who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis, and in the opinion of the Principal Investigator.
* Female participants (if of child-bearing potential and sexually active) who agree to use a medically acceptable and effective birth control method throughout the study and for 30 days following the end of the study
* Male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method from the first dose and for 90 days following last dose of study drug. Male participants must refrain from donating sperm for the same period.

Exclusion Criteria:

* Subject history, which includes: any cardiovascular disease or disorder; asthma, chronic obstructive lung disease, or any use of an inhaler prescribed for wheezing or bronchospasm must be excluded; sleep apnea; acute narrow-angle glaucoma; any neurological, gastrointestinal, hepatic, renal, hematologic, endocrine and/or metabolic disease or disorder; psychiatric illness or mental disorder except for short term situational anxiety or depression of < 2 years duration; any substance abuse or addiction within the last 2 years; pregnancy within the past 6 months.
* Subjects who have taken prescription or nonprescription medication within 7 days of Visit 2.
* Subjects who have had an acute illness within the last 7 days of Visit 2.
* Subjects who have a history of HIV positivity.
* Subjects who test positive for alcohol or have a positive urine drug screen.
* Subjects who have a history of allergy or intolerance to loxapine or amoxapine.
* Subjects who have a history of allergy or intolerance to lorazepam or any other benzodiazepine.
* Subjects who have a history of allergy or intolerance to polyethylene glycol, propylene glycol, or benzyl alcohol
* Female subjects who have a positive pregnancy test at screening or at admission to Visit 2, or are breastfeeding.
* Subjects who have received an investigational drug within 30 days prior to the Screening Visit.
* Subjects who have any other disease(s), by history, physical examination, or laboratory abnormalities that, in the investigator's opinion, presents undue risk to the subject or may confound the interpretation of study results.
* Subjects who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving lorazepam or ADASUVE.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall R Stoltz, MD, Principal Investigator — Medical Director, Covance-Evansville, Evansville, IN 47710
Locations (1):
- Covance-Evansville, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Result] Spyker DA, Cassella JV, Stoltz RR, Yeung PP. Inhaled loxapine and intramuscular lorazepam in healthy volunteers: a randomized placebo-controlled drug-drug interaction study. Pharmacol Res Perspect. 2015 Dec 17;3(6):e00194. doi: 10.1002/prp2.194. eCollection 2015 Dec. PMID 27022468

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label (Lorazepam 1 mg + Inhaled Loxapine 10 mg): Inhaled Staccato loxapine 10 mg + IM lorazepam 1 mg
  Lorazepam 1 mg IM: Lorazepam 1 mg intramuscular
  Inhaled loxapine 10 mg: Inhaled Staccato loxapine 10 mg
Period: Overall Study
Arm/Group | Open Label (Lorazepam 1 mg + Inhaled Loxapine 10 mg) | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BCA | Treatment Sequence BAC | Treatment Sequence CAB | Treatment Sequence CBA
Started | 4 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 4 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Open Label Subjects: Open label portion of study
- All Crossover Subjects: All 6 crossover treatment sequences
- Total: Total of all reporting groups
Arm/Group | Open Label Subjects | All Crossover Subjects | Total
Number analyzed (Participants) | 4 | 18 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 18 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.68) | 30.4 (9.46) | 30.8 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 2 | 11 | 13
Region of Enrollment [Number; unit: participants]
  United States | 4 | 18 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Level of Sedation for Lorazepam 1 mg IM + ADASUVE 10 mg
Description: Determine the maximum level of sedation for Lorazepam 1 mg IM + ADASUVE 10 mg based on the 100 mm Visual Analog Scale (VAS) ranging from (0=sleepy to 100=wide awake)
Time Frame: 24 hours
Population: Open label population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Open Label Group: Lorazepam 1 mg IM + Inhaled loxapine 10 mg
Arm/Group | Open Label Group
Number analyzed (Participants) | 4
units on a scale | 12.3 (6.65)

2. Primary Outcome: Relative Pharmacodynamic Effect on Respiration Rate for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Mean ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for respiration rate following administration of Lorazepam+Loxapine compared to the same measure following each control drug given alone (Lorazepam, Loxapine)
Time Frame: 24 hours
Population: Pharmacodynamics Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Groups:
- Lorazepam+Loxapine / Lorazepam: Lorazepam 1 mg IM + Inhaled Staccato Loxapine 10 mg compared to Lorazepam 1 mg IM
- Lorazepam+Loxapine / Loxapine: Lorazepam 1 mg IM + Inhaled Staccato Loxapine 10 mg compared to Inhaled Loxapine 10 mg
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 94.3 [91.5 to 97.3] | 97.3 [94.3 to 100]

3. Secondary Outcome: Relative Pharmacodynamic Effect on Systolic Blood Pressure for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for systolic blood pressure following administration of Lorazepam+Loxapine compared to the same measure following each control drug (Lorazepam, Loxapine) given alone
Time Frame: 24 hours
Population: Pharmacodynamics Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 100 [97.8 to 103] | 102 [97.8 to 105]

4. Secondary Outcome: Relative Pharmacodynamic Effect on Sedation for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for sedation based on a 100 mm Visual Analog Scale (VAS) ranging from (0=sleepy to 100=wide awake) following administration of Lorazepam+Loxapine compared to the same measure following each control drug given alone (Lorazepam, Loxapine)
Time Frame: 24 hours
Population: Pharmacodynamics Population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 41.7 [33.8 to 51.5] | 95.7 [77.6 to 118]

5. Secondary Outcome: Relative Pharmacodynamic Effect on Pulse Oximetry for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for pulse oximetry following administration of Lorazepam+Loxapine compared to the same measure following each control drug (Lorazepam, Loxapine) given alone
Time Frame: 24 hours
Population: Pharmacodynamic population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 99.7 [99.4 to 100.1] | 100.3 [100.0 to 100.6]

6. Secondary Outcome: Relative Pharmacodynamic Effect on Heart Rate for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for heart rate following administration of Lorazepam+Loxapine compared to the same measure following each control drug (Lorazepam, Loxapine) given alone
Time Frame: 24 hours
Population: Pharmacodynamic population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 96.9 [91.4 to 102.7] | 99.7 [94.0 to 105.7]

7. Secondary Outcome: Relative Pharmacodynamic Effect on Diastolic Blood Pressure for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for diastolic blood pressure following administration of Lorazepam+Loxapine compared to the same measure following each control drug (Lorazepam, Loxapine) given alone
Time Frame: 24 hours
Population: Pharmacodynamic population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 101.8 [98.0 to 105.7] | 100.3 [96.6 to 104.2]

8. Secondary Outcome: Relative Pharmacodynamic Effect on Cogscreen Pathfinder Response for Combined vs Individual (Lorazepam, Loxapine)
Description: LS Means ratio (90% CI) of the area under the curve for 0 to 24 hours (AUC 0-24) for Cogscreen Pathfinder Response following administration of Lorazepam+Loxapine compared to the same measure following each control drug (Lorazepam, Loxapine) given alone
Time Frame: 24 hours
Population: Pharmacodynamic population
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of effect on control drug
Arm/Group | Lorazepam+Loxapine / Lorazepam | Lorazepam+Loxapine / Loxapine
Number analyzed (Participants) | 18 | 18
percentage of effect on control drug | 134 [122 to 147] | 133 [121 to 146]

ADVERSE EVENTS:
Time Frame: From time of first study treatment to 30 days after the last study treatment
Description: Adverse events reported to the investigator by telephone report, by historical report at the follow-up visit, or to study personnel during the follow-up assessment, regardless of treatment group (if known) or suspected causal relationship to study drug, were recorded on the AE CRF. AEs were collected pre-dose, 15, 30, 45, 60, 75, 90 & 105 min; 2, 3, 4, 5, 6, 7, 8, 9 12 and 24 hours.
Groups:
- Lorazepam 1 mg IM: Lorazepam 1 mg IM + Inhaled placebo
  Lorazepam 1 mg IM: Lorazepam 1 mg intramuscular
  Inhaled Placebo: Inhaler with no drug in it to mimic the ADASUVE inhaler
- Lorazepam 1 mg IM + Inhaled Loxapine 10 mg: Lorazepam 1 mg IM + Inhaled Staccato loxapine 10 mg
  Lorazepam 1 mg IM: Lorazepam 1 mg intramuscular
  Inhaled loxapine 10 mg: Inhaled Staccato loxapine 10 mg
- Inhaled Loxapine 10 mg: Inhaled Staccato loxapine 10 mg + IM placebo
  Inhaled loxapine 10 mg: Inhaled Staccato loxapine 10 mg
  Placebo IM: intramuscular placebo to mimic lorazepam 1 mg IM
Arm/Group | Open Label (Lorazepam 1 mg + Inhaled Loxapine 10 mg) | Lorazepam 1 mg IM | Lorazepam 1 mg IM + Inhaled Loxapine 10 mg | Inhaled Loxapine 10 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/4 | 0/18 | 0/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (Lorazepam 1 mg + Inhaled Loxapine 10 mg) (N=4) | Lorazepam 1 mg IM (N=18) | Lorazepam 1 mg IM + Inhaled Loxapine 10 mg (N=18) | Inhaled Loxapine 10 mg (N=18)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The 1-mg IM lorazepam dose used in this study was lower than that used in some previous studies assessing the effects of concomitant administration of antipsychotics with up to 2-mg lorazepam for the treatment of agitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less